CLINICAL TRIAL: NCT00032045
Title: An Open-label Study Of MDX-010 In Combination With gp100 Peptides Emulsified With Montanide ISA 51 In The Treatment Of Patients With Stage IV Melanoma
Brief Title: Vaccine Therapy and Monoclonal Antibody Therapy in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069251; NCI-02-C-0106H; NCI-5743; NCT00029549 (obsolete NCT alias)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2003-03

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: iris melanoma; ciliary body and choroid melanoma, small size; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; recurrent intraocular melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — incomplete Freund's adjuvant; Ipilimumab

INTERVENTIONS:
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: ipilimumab

SUMMARY:
RATIONALE: Vaccines made from peptides may make the body build an immune response to kill tumor cells. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining vaccine therapy with a monoclonal antibody may cause a stronger immune response and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining vaccine therapy with monoclonal antibody therapy in treating patients who have stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical response in patients with stage IV melanoma when treated with anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody combined with gp100:209-217 and gp100:280-288 peptides emulsified in Montanide ISA-51.
* Determine a safety and adverse event profile of this regimen in these patients.
* Determine improved immunologic response in patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody IV over 90 minutes immediately followed by gp100:209-217 and gp100:280-288 peptides emulsified in Montanide ISA-51 subcutaneously on days 1, 22, 43, and 64. Treatment repeats every 12 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 weeks, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 68 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV melanoma

  * Mucosal or ocular melanoma allowed
* Clinically evaluable disease
* HLA-A*0201 positive

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 6 months

Hematopoietic:

* WBC at least 2,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL
* Hematocrit at least 30%

Hepatic:

* AST no greater than 3 times upper limit of normal (ULN)
* Bilirubin no greater than ULN (less than 3.0 mg/dL in patients with Gilbert's syndrome)
* Hepatitis B surface antigen negative
* Hepatitis C antibody nonreactive

Renal:

* Creatinine less than 2.0 mg/dL

Immunologic:

* Antinuclear antibody negative
* Thyroglobulin antibody normal
* Rheumatoid factor normal
* HIV negative
* No prior autoimmune disease (including uveitis and autoimmune inflammatory eye disease)
* No active infection
* No hypersensitivity to Montanide ISA-51

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* No other underlying medical condition that would preclude study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior immunotherapy for melanoma and recovered
* No prior gp100 peptides
* No prior anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody

Chemotherapy:

* At least 3 weeks since prior chemotherapy for melanoma and recovered
* No concurrent chemotherapy

Endocrine therapy:

* At least 3 weeks since prior hormonal therapy for melanoma and recovered
* At least 4 weeks since prior systemic or topical corticosteroids
* No concurrent topical or systemic corticosteroids

Radiotherapy:

* At least 3 weeks since prior radiotherapy for melanoma and recovered

Surgery:

* Not specified

Other:

* No other concurrent immunosuppressive agents (e.g., cyclosporine and its analog)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-01; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Background] Maker AV, Attia P, Rosenberg SA. Analysis of the cellular mechanism of antitumor responses and autoimmunity in patients treated with CTLA-4 blockade. J Immunol. 2005 Dec 1;175(11):7746-54. doi: 10.4049/jimmunol.175.11.7746. PMID 16301685
- [Background] Maker AV, Phan GQ, Attia P, Yang JC, Sherry RM, Topalian SL, Kammula US, Royal RE, Haworth LR, Levy C, Kleiner D, Mavroukakis SA, Yellin M, Rosenberg SA. Tumor regression and autoimmunity in patients treated with cytotoxic T lymphocyte-associated antigen 4 blockade and interleukin 2: a phase I/II study. Ann Surg Oncol. 2005 Dec;12(12):1005-16. doi: 10.1245/ASO.2005.03.536. Epub 2005 Oct 21. PMID 16283570
- [Result] Attia P, Phan GQ, Maker AV, Robinson MR, Quezado MM, Yang JC, Sherry RM, Topalian SL, Kammula US, Royal RE, Restifo NP, Haworth LR, Levy C, Mavroukakis SA, Nichol G, Yellin MJ, Rosenberg SA. Autoimmunity correlates with tumor regression in patients with metastatic melanoma treated with anti-cytotoxic T-lymphocyte antigen-4. J Clin Oncol. 2005 Sep 1;23(25):6043-53. doi: 10.1200/JCO.2005.06.205. Epub 2005 Aug 8. PMID 16087944
- [Result] Phan GQ, Yang JC, Sherry RM, Hwu P, Topalian SL, Schwartzentruber DJ, Restifo NP, Haworth LR, Seipp CA, Freezer LJ, Morton KE, Mavroukakis SA, Duray PH, Steinberg SM, Allison JP, Davis TA, Rosenberg SA. Cancer regression and autoimmunity induced by cytotoxic T lymphocyte-associated antigen 4 blockade in patients with metastatic melanoma. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8372-7. doi: 10.1073/pnas.1533209100. Epub 2003 Jun 25. PMID 12826605
- [Derived] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295